CLINICAL TRIAL: NCT00182624
Title: Comprehensive Prostate MRI for the Evaluation of Prostate Cancer at 3.0T: A Pilot Study
Brief Title: Magnetic Resonance Imaging to Evaluate Prostate Cancer
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040109; 04-CC-0109; NCT00076908 (obsolete NCT alias)
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-09-06

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; Magnetic Resonance Imaging; Spectroscopy
MeSH Terms: conditions — Prostatic Neoplasms

SUMMARY:
This study will determine whether scanning the prostate using special magnetic resonance imaging (MRI) techniques can detect prostate cancers with greater accuracy than other methods. MRI uses a strong magnet and radio waves to produce images of body tissues. Unlike many cancers, prostate cancer is difficult to see on most imaging studies like x-rays, computed tomography (CT) scans, and conventional MRI scans. This study will use a magnet twice as strong as the magnets commonly used in MRI tests.

Patients 18 years of age and older with prostate cancer confirmed by prostate biopsy may be eligible for this study. Candidates are screened with a medical history, physical examination, and review of pathology reports.

Participants undergo MRI of the prostate and possibly a biopsy of the prostate gland, as follows:

Prostate MRI

Before coming to the NIH Clinical Center for the biopsy, patients take a Fleets enema to empty the rectum of fecal matter. For the MRI, an endorectal coil (a tube containing a specially designed antenna) is placed in the rectum, which is just behind the prostate. The coil increases the amount of signal received by the MRI unit. Additional coils may be wrapped around the pelvis to further improve the quality of the scan. The patient lies on a stretcher that moves into the scanner. A catheter (plastic tube) is placed in an arm vein for injection of a contrast agent called gadolinium, which brightens the images. Patients may also be asked to breathe an oxygen-rich gas through a mask during the scan to test the use of oxygen as a contrast agent in MRI. Patients may be asked to repeat the MRI to test the reproducibility of the procedure. The repeat test is optional.

Prostate Biopsy

Depending on the MRI findings, patients may be asked to undergo a prostate biopsy to obtain a sample of tumor tissue. The tissue is obtained with a needle placed through the rectum. Medicines may be used to reduce pain during the biopsy and to reduce the chance of infection.

DETAILED DESCRIPTION:
Progress in effective local therapy of prostate cancer has been stymied by the lack of an imaging technique capable of reliably identifying the location of cancer within the prostate. Magnetic Resonance Imaging is a promising candidate for imaging the prostate because of its high soft tissue contrast, multiplanar capabilities, and the potential for providing unique biologic information not available with other modalities. In addition to conventional T2-weighted imaging MRI techniques that provide unique biologic information include MR spectroscopy, diffusion weighted MRI, dynamic enhanced MRI and hypoxia imaging. All have shown promise in imaging tumors at a magnetic field strength of 1.5 Tesla but all have been limited by sensitivity. Since MR signal is proportional to magnetic field strength, 3.0 Tesla clinical systems potentially could improve overall diagnostic accuracy. A comprehensive imaging package which incorporates all these techniques to study prostate cancer on a state-of-the-art 3.0 Tesla magnet has not yet been developed.

In this pilot study we seek to develop and evaluate a comprehensive prostate MR exam at 3.0 Tesla. Patients with biopsy proven prostate cancer will undergo an MRI with endorectal and surface phased array coils which will include conventional sequences, MR spectroscopy, Diffusion weighted MRI, Dynamic enhanced MR and Hypoxia imaging. In the development phase of this trial (30 patients), the robustness of the techniques and test-retest reproducibility will be evaluated. In the second phase, the comprehensive prostate MRI exam will be validated against the results of prostate biopsy (50 patients). The expected accrual period is two years. We hope that this method will offer prostate cancer patients a more accurate method of localizing their prostate cancer than is now possible which should improve outcomes and minimize complications of treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recent transrectal biopsy of the prostate gland in which at least sextant biopsies were obtained. Knowledge of the location of each specimen is required for inclusion.

Age greater than or equal to18 years.

ECOG performance status of 0 or 1.

Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

EXCLUSION CRITERIA:

Patients with contraindication to endorectal coil placement.

* Bleeding disorder documented by history.
* Severe immunocompromise documented by history.
* PT/PTT greater than 1.5 times the upper limit of normal.
* Platelets less than 50K.
* Artificial heart valve.
* Severe hemorrhoids.
* Surgically absent rectum.

Patients with contraindications to MRI.

* Patients weighing greater than 136 kg (weight limit for scanner table).
* Patients with pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices not compatible with MRI.

Patients with contraindications to prostate biopsy.

* See above contraindications for endorectal coil placement.
* Previous severe adverse event with prostatic biopsies.

Patients with distant metastatic disease.

Patients with a prior history of pelvic or prostate radiotherapy.

Patient with a prior history of androgen ablative hormonal therapy (orchiectomy, LHRH analogues, anti-androgens).

Cognitively impaired patients who cannot give informed consent.

Other medical conditions deemed by the PI or associates to make the patient ineligible for protocol procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-02-02; Study Completion 2007-09-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gibbs P, Tozer DJ, Liney GP, Turnbull LW. Comparison of quantitative T2 mapping and diffusion-weighted imaging in the normal and pathologic prostate. Magn Reson Med. 2001 Dec;46(6):1054-8. doi: 10.1002/mrm.1298. PMID 11746568